CLINICAL TRIAL: NCT04867980
Title: Randomized, Double-Blind, Double-Dummy, Placebo- and Positive Controlled, 4-Way Crossover Study to Assess the Effect of Single-Dose ACP-196 on the QTc Interval in Healthy Adult Subjects
Brief Title: A Study to Evaluate the Effect of ACP-196 on the Heart Rate-corrected QT Interval in Healthy Adult Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Acerta Pharma BV (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ACE-HV-005
Record Dates: First submitted 2021-04-28; First posted 2021-04-30 (Actual); Last update posted 2021-04-30 (Actual); Status verified 2021-04

CONDITIONS: Healthy Volunteers
Keywords: ACE-HV-005; ACP-196; Healthy participants; Volunteers; Adults; QTc Interval; Pharmacokinetics; PK
MeSH Terms: interventions — acalabrutinib; Moxifloxacin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- ABCD (Experimental): Participant will receive a single oral dose of 4 study treatments with the sequences of ABCD. The washout period will be >= 5 days between each dose.
  Interventions: Drug: ACP-196; Drug: Moxifloxacin 400 mg; Drug: Placebo
- BDAC (Experimental): Participant will receive a single oral dose of 4 study treatments with the sequences of BDAC. The washout period will be >= 5 days between each dose.
  Interventions: Drug: ACP-196; Drug: Moxifloxacin 400 mg; Drug: Placebo
- CADB (Experimental): Participant will receive a single oral dose of 4 study treatments with the sequences of CADB. The washout period will be >= 5 days between each dose.
  Interventions: Drug: ACP-196; Drug: Moxifloxacin 400 mg; Drug: Placebo
- DCBA (Experimental): Participant will receive a single oral dose of 4 study treatments with the sequences of DCBA. The washout period will be >= 5 days between each dose.
  Interventions: Drug: ACP-196; Drug: Moxifloxacin 400 mg; Drug: Placebo

INTERVENTIONS:
Drug: ACP-196 — Participants will receive a single oral dose of 100 mg ACP-196 (1 x 100 mg capsule) on Day 1 (Treatment A) and 400 mg ACP-196 (4 x 100 mg capsules) on Day 1 (Treatment B) according to the randomization scheme.
  Other Names: Acalabrutinib
Drug: Moxifloxacin 400 mg — Participants will receive a single oral dose of 400 mg moxifloxacin (1 x 400 mg tablet) on Day 1 (Treatment C) according to the randomization scheme.
Drug: Placebo — Participants will receive a single oral dose of ACP-196 matching placebo (4 x 100 mg matching placebo capsules) and moxifloxacin matching placebo (1 x 400 mg matching placebo tablet) on Day 1 (Treatment D) according to the randomization scheme.

SUMMARY:
This study is to evaluate the effects of single therapeutic and supratherapeutic oral doses of ACP-196 on the heart rate-corrected QT interval using Fridericia's formula (QTcF).

DETAILED DESCRIPTION:
This is a single-dose, randomized, double-blind, double-dummy, placebo- and positive-controlled, 4-period, balanced crossover study under fasting conditions. Participants will be randomized to 1 of 4 treatment sequences: ABCD, BDAC, CADB, or DCBA. On 4 different occasions (4 periods), each participant will receive Treatment A (a single therapeutic oral dose of 100 mg ACP-196), Treatment B (a single supratherapeutic oral dose of 400 mg ACP-196), Treatment C (a single oral dose of 400 mg moxifloxacin) or Treatment D (a single oral dose of ACP-196 and moxifloxacin matching placebos) according to a randomization scheme. The washout period will be >= 5 days between each dose. The clinic attempted to contact participants using their standard procedures approximately 14 days after the last study drug (or placebo) administration to determine if any adverse events (AEs) had occurred since the last dose of study drug(s). An adverse event is any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship.

ELIGIBILITY:
Inclusion Criteria:

* Continuous non-smoker participant who has not used nicotine-containing products for >= 3 months before the first dose
* Have body mass index of >= 18.0 and <= 32.0 kg/m^2 at screening
* Medically healthy with no clinically significant medical history, physical examination, laboratory profiles, vital signs, or electrocardiograms (ECGs), as deemed by the principal investigator (PI)
* No clinically significant history or presence of ECG findings as judged by the PI or qualified designee at screening and each check-in, including each criterion as: 1) Normal sinus rhythm (heart rate between 50 and 100 beats per minute [bpm]), 2) QTcF interval ≤ 450 milliseconds (msec), 3) QRS interval ≤ 110 msec, and 4) PR interval ≤ 220 msec
* Women participants must be of non-childbearing status
* Women participants must have negative serum pregnancy test
* ability to swallow multiple capsules and/or tablets using size 0 blank capsules (up to a maximum of 5 capsules per participant)
* Male participants must be willing to use protocol specified contraception methods

Exclusion Criteria:

* Participant is mentally or legally incapacitated or has significant emotional problems at the time of the screening visit or expected during the conduct of the study
* History of any illness that, in the opinion of the PI, might confound the results of the study or poses an additional risk to the subject by their participation in the study
* Presence of any clinically significant, ongoing systemic bacterial, fungal, or viral infections (including upper respiratory tract infections, but excluding localized cutaneous fungal infections), in the opinion of the PI
* History of any major surgical procedure within 30 days before the first dose of study drug
* History or presence of alcoholism or drug abuse within the past 2 years before screening
* Any clinically significant condition that may affect ACP-196 absorption in the opinion of the PI, including gastric restrictions and bariatric surgery (eg, gastric bypass).
* Allergy to band-aids, adhesive dressing, or medical tape
* History or presence of clinically significant thyroid disease
* Prior exposure to Bruton's tyrosine kinase inhibitors (eg, ACP-196, ibrutinib) within 3 months before the first dose of study drug
* Positive urine cotinine at screening
* Positive urine drug or alcohol results at screening or each check-in
* Positive for human immunodeficiency virus (HIV), hepatitis B surface antigen (HBsAg), or hepatitis C virus (HCV) at screening
* Seated blood pressure is less than 90/40 mmHg or greater than 140/90 mmHg at screening
* Seated heart rate is lower than 50 bpm or higher than 99 bpm at screening
* Unable to refrain from or anticipates the use of protocol defined medications for 28 days before the first dose of study drug and throughout the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2016-04-01 (Actual); Primary Completion 2016-05-09 (Actual); Study Completion 2016-05-09 (Actual)

PRIMARY OUTCOMES:
The QTcF Change From Baseline at Postdose Timepoints (dQTcF) | 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 8, 12, and 24 hours postdose in each period

SECONDARY OUTCOMES:
Change in Time-matched QTcF Interval Following Moxifloxicin Administration Compared With Matching Placebo | 1, 2, 3, and 4 hour post moxifloxicin dose in each period
Change From Baseline in Heart Rate at Postdose Time Points | 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 8, 12, and 24 hours postdose in each period
Change From Baseline in PR Interval at Postdose Time Points | 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 8, 12, and 24 hours postdose in each period
Change From Baseline in RR Interval at Postdose Time Points | 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 8, 12, and 24 hours postdose in each period
Change From Baseline in QRS Interval at Postdose Time Points | 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 8, 12, and 24 hours postdose in each period
Change From Baseline in QT Interval at Postdose Time Points | 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 8, 12, and 24 hours postdose in each period
Number of Participants With Nonspecific T Waves Abnormality at Postdose Time Points | 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 8, 12, and 24 hours postdose in each period
Number of Participants With Nonspecific U Waves Abnormality at Postdose Time Points | 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 8, 12, and 24 hours postdose in each period
Area Under the Plasma Concentration-time Curve From Time 0 to Time of Last Measurable Concentration (AUC0-last) of ACP-196 | -0.5, 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 8, 12, and 24 hours postdose in each period
Area Under the Plasma Concentration-time Curve From Time 0 to Infinity (AUC0-inf) of ACP-196 | -0.5, 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 8, 12, and 24 hours postdose in each period
Percent of AUC0-inf Extrapolated (AUC%extrap) of ACP-196 | -0.5, 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 8, 12, and 24 hours postdose in each period
Maximum Measured Plasma Concentration (Cmax) of ACP-196 | -0.5, 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 8, 12, and 24 hours postdose in each period
Time of the Maximum Measured Plasma Concentration (Tmax) of ACP-196 | -0.5, 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 8, 12, and 24 hours postdose in each period
Apparent Terminal Elimination Rate Constant (λz) of ACP-196 | -0.5, 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 8, 12, and 24 hours postdose in each period
Apparent Terminal Elimination Half-life ( t½) of ACP-196 | -0.5, 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 8, 12, and 24 hours postdose in each period
Apparent Total Plasma Clearance (CL/F) of ACP-196 | -0.5, 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 8, 12, and 24 hours postdose in each period
Incidence of Treatment-emergent Adverse Events (TEAEs) and Treatment-emergent Serious AEs (TESAEs) | From Day 1 through 14 days after the last dose of study drug of the last period (approximately 1 month and 8 days)
Incidence of Abnormal Clinical Laboratory Parameters Reported as TEAEs | From Day 1 through 24 hours after the last dose of study drug of the last period (approximately 1 month and 8 days)
Incidence of Abnormal Vital Signs and Physical Examinations Reported as TEAEs | From Day 1 through 24 hours after the last dose of study drug of the last period (approximately 1 month and 8 days)
Incidence of Abnormal ECGs Reported as TEAEs | From Day 1 through 24 hours after the last dose of study drug of the last period (approximately 1 month and 8 days)

CONTACTS AND LOCATIONS:
Overall Officials: Priti Patel, MD, Study Director — Acerta Clinical Trials
Locations (1):
- Celerion, Tempe, Arizona, United States

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal. All request will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
  Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the de-identified individual patient-level data in an approved sponsored tool. Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home